CLINICAL TRIAL: NCT02532556
Title: Electrical Stimulation of the Muscle Pumps of the Leg
Acronym: Muscle Pump
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Triple | Purpose: Basic Science
Other Study IDs: 15IC2528
Record Dates: First submitted 2015-08-10; First posted 2015-08-25 (Estimated); Results first posted 2020-11-27 (Actual); Last update posted 2020-11-27 (Actual); Status verified 2020-11

CONDITIONS: Haemodynamic Physiology
Keywords: Haemodynamic physiology
MeSH Terms: interventions — Electric Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- 1 (Experimental): Stimulation of muscle in this order: vastus medials, rectus femoris, vastus lateralis, tibialis anterior, peroneus longus, medial head gastrocnemius, lateral head gastrocnemius
  Interventions: Device: Electrical stimulation (Digitimer)
- 2 (Experimental): Stimulation of muscle in this order: rectus femoris, vastus lateralis, tibialis anterior, peroneus longus, medial head gastrocnemius, lateral head gastrocnemius, vastus medials
  Interventions: Device: Electrical stimulation (Digitimer)
- 3 (Experimental): Stimulation of muscle in this order: vastus lateralis, tibialis anterior, peroneus longus, medial head gastrocnemius, lateral head gastrocnemius, vastus medials, rectus femoris
  Interventions: Device: Electrical stimulation (Digitimer)
- 4 (Experimental): Stimulation of muscle in this order: tibialis anterior, peroneus longus, and the medial head gastrocnemius, lateral head gastrocnemius, vastus medials, rectus femoris, vastus lateralis
  Interventions: Device: Electrical stimulation (Digitimer)
- 5 (Experimental): Stimulation of muscle in this order: peroneus longus, medial head gastrocnemius, lateral head gastrocnemius, vastus medials, rectus femoris, vastus lateralis, tibialis anterior
  Interventions: Device: Electrical stimulation (Digitimer)
- 6 (Experimental): Stimulation of muscle in this order: medial head gastrocnemius, lateral head gastrocnemius, vastus medials, rectus femoris, vastus lateralis, tibialis anterior, peroneus longus
  Interventions: Device: Electrical stimulation (Digitimer)
- 7 (Experimental): Stimulation of muscle in this order: lateral head gastrocnemius, vastus medials, rectus femoris, vastus lateralis, tibialis anterior, peroneus longus, medial head gastrocnemius,
  Interventions: Device: Electrical stimulation (Digitimer)

INTERVENTIONS:
Device: Electrical stimulation (Digitimer) — Stimulation with Digitimer (DS7A HV, Digitimer Ltd, UK) over motor point of muscle in protocol. 1Hz, pulse duration 1ms, maximum compliance voltage 200V. Current set to twice motor threshold

SUMMARY:
The most efficient way of electrically stimulating the calf muscles has not been identified. The investigators aim to investigate this using a matrix of electrical parameters, and measuring the outcome with vascular ultrasound of the leg.

DETAILED DESCRIPTION:
Blood is aided on its journey to the heart by the action of the muscles of the legs. Muscle contraction squeezes the deep veins of the leg and pushes blood upwards, back towards the heart. In immobilised patients, or those with blood vessel problems, the pumping process can be helped by machines that either squeeze or shock the muscles of the calf (e.g. intermittent pneumatic compression, electrical stimulating devices). Many are licensed for medical use, and some are common place in hospitals and outpatient departments.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Current good health

Exclusion Criteria:

* History of cardiovascular disease
* Ankle Brachial Pressure Index <0.9
* Venous reflux>0.5s
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2015-05; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alun Davies, Principal Investigator — Imperial College London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Evans DR, Williams KJ, Strutton PH, Davies AH. The comparative hemodynamic efficacy of lower limb muscles using transcutaneous electrical stimulation. J Vasc Surg Venous Lymphat Disord. 2016 Apr;4(2):206-14. doi: 10.1016/j.jvsv.2015.10.009. Epub 2016 Jan 12. PMID 26993869

RESULTS

PARTICIPANT FLOW:
Groups:
- Electrical Muscle Stimulation Participants: All participants for electrical stimulation of respective muscles (tibialis anterior, peroneus longus, gastrocnemius, vastus lateralis, rectus femoris, vastus medialis)
Period: Overall Study
Arm/Group | Electrical Muscle Stimulation Participants
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Electrical Muscle Stimulation Participants
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 23.1 (3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 5
Region of Enrollment [Number; unit: participants]
  United Kingdom | 12
Body mass index [Mean (Standard Deviation); unit: kg/m^2] | 23.1 (3)

OUTCOME MEASURES:

1. Primary Outcome: Venous Haemodynamic Measurements (Volume Flow Rate)
Description: Measurement by ultrasound, in right femoral vein. Flow rate (ml/min).
Time Frame: Baseline compared to that after 10-mins stimulation (2-mins to take measurements)
Population: Muscle stimulated
Measure: Median (Standard Deviation); unit: ml/min
Arm/Group | Vastus Lateralis | Rectus Femoris | Vastus Medialis | Gastrocnemius (Medial) | Gastrocnemius (Lateral) | Tibialis Anterior | Peroneus Longus
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 12 | 12 | 12
ml/min
  Baseline | 119 (67) | 158 (123) | 158 (134) | 144 (100) | 161 (168) | 164 (66) | 139 (135)
  Stimulation | 148 (97) | 158 (123) | 150 (125) | 178 (120) | 114 (205) | 153 (171) | 149 (113)
Statistical Analysis 1: Comparison: Gastrocnemius (Medial); Test type: Superiority; p < 0.05, Wilcoxan signed-rank test

2. Primary Outcome: Venous Haemodynamic Measurements (Time Averaged Maximum Velocity)
Description: Measurement by ultrasound, in right femoral vein. Time averaged maximum velocity (cm/s).
Time Frame: Baseline compared to that after 10-mins stimulation (2-mins to take measurements)
Population: Muscle stimulated
Measure: Median (Standard Deviation); unit: cm/s
Arm/Group | Vastus Lateralis | Rectus Femoris | Vastus Medialis | Gastrocnemius (Medial) | Gastrocnemius (Lateral) | Tibialis Anterior | Peroneus Longus
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 12 | 12 | 12
cm/s
  Baseline | 8.2 (10) | 8.8 (14) | 11.3 (10) | 8.5 (12) | 7.5 (12) | 11.3 (13) | 13.4 (14)
  Stimulation | 8.2 (15) | 10.6 (10) | 10.9 (8) | 11.6 (19) | 10.5 (11) | 12 (9) | 10.8 (17)
Statistical Analysis 1: Comparison: Gastrocnemius (Medial); Test type: Superiority; p < 0.05, Wilcoxan signed-rank test

3. Secondary Outcome: Pain Grading on Stimulation
Description: Visual analogue scale (0-minimum pain, to 100-maximum pain)
Time Frame: During stimulation (10-mins each muscle)
Population: Muscle stimulated
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Vastus Lateralis | Rectus Femoris | Vastus Medialis | Gastrocnemius (Medial) | Gastrocnemius (Lateral) | Tibialis Anterior | Peroneus Longus
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 12 | 12 | 12
scores on a scale | 15 (1) | 66.3 (1) | 21.3 (1) | 28.8 (1) | 31.3 (1) | 21.3 (1) | 30 (1)

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Electrical Muscle Stimulation Participants
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes